CLINICAL TRIAL: NCT00881192
Title: Perioperative IABP in CABG Operations in Patients With Severely Depressed Left Ventricular Function: a Randomized, Controlled Trial
Brief Title: Perioperative Intra-Aortic Balloon Pump (IABP) in Coronary Artery Bypass Grafting (CABG) Operations in Patients With Severely Depressed Left Ventricular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Marco Ranucci, Anesthesia and Reanimation Clinical Research Director, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IABPCABG
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Coronary Artery Disease; Coronary Artery Bypass Grafting
Keywords: CABG; coronary surgery; intra-aortic balloon pump; CABG operation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No preoperative IABP; if needed, postoperative IABP placement
- IABP (Active Comparator): Preoperative IABP placement
  Interventions: Procedure: IABP

INTERVENTIONS:
Procedure: IABP — preoperative IABP placement
  Arms: IABP

SUMMARY:
Since its first introduction in humans in 1962, Intra-Aortic Balloon Pump (IABP) is now the most commonly used therapeutic option to support failing heart in cardiac surgery. The main effects of IABP are an increase in diastolic blood pressure and therefore an improvement in coronary perfusion and a reduction of ventricular after load, thus increasing stroke volume and cardiac output. IABP-related complications include limb ischemia, bleeding at the site of IABP insertion, infection, and aortic dissection.

IABP could be used preoperatively, intraoperatively, or postoperatively. However, despite the wide use of the device, the optimal timing and use of IABP in high-risk patients undergoing cardiac surgery remains controversial. Time of insertion has been showed to affect hospital mortality, ranging from 18.8% to 19.6% for preoperative insertion, from 27.6% to 32.3% for intraoperative insertion, and from 39% to 40.5% for postoperative insertion. Several studies, randomized and non-randomized, have been conducted to address the impact of preoperative use of IABP on the outcome, each study including a relative small number of patients. In an effort to increase the strength of the results, two meta-analysis have been conducted and published in 2008. The objectives of both were to assess the effect on mortality and morbidity of using IABP preoperatively in high-risk patients undergoing coronary artery bypass grafting (CABG). Surprisingly, the meta-analysis from Field and co-workers was conducted on four randomized controlled trials (for a total of 193 patients included) published by the same author from the same institution, making the results not conclusive although favourable toward a beneficial effect of the preoperative use of IABP. Moreover, two of the randomized trials conducted by Christenson and co-workers and included in the above mentioned meta-analysis, were excluded from the meta-analysis from Dyub and co-workers because considered duplicates. Unfortunately, one study by Christenson and co-workers and included in the meta-analysis from Dyub was conducted on off-pump surgery, introducing another bias in the criteria of eligibility.

At present it is unclear whether the preoperative use of IABP in high-risk coronary patients scheduled for CABG operations leads to a better outcome. The experimental hypothesis of the present randomized, controlled trial (RCT) is that the placement of IABP immediately before beginning the surgical procedure induces a reduction of major morbidity after the operation.

DETAILED DESCRIPTION:
RCT including patients scheduled for elective CABG surgery (with or without associated procedures) and having a left ventricular ejection fraction < 0.35. Exclusion criteria: age < 18 years, no patient's consent, contra-indications to the use of IABP (severe peripheral arteropathy; endovascular abdominal aortic prostheses).

Patients will be randomly allocated to either a control group or a treatment group. Patients in the control group will not receive an IABP preoperatively, and patients in the treatment arm will receive an IABP positioned immediately after the induction of anesthesia and before beginning surgery.

Randomization will be performed the day before the operation. Primary endpoint: reduction of major morbidity rate (defined as either prolonged (> 48 hours) mechanical ventilation, acute renal failure, mediastinitis, surgical revision, stroke).

Secondary endpoint: reduction in inotropic drug use, shortening of mechanical ventilation and ICU stay.

Interim analyses and stopping rules: interim analyses will be done at half (80 patients)and 2/3 (106 patients) of recruitment. The trial could be prematurely stopped in case of a difference in the primary endpoint reaching a P value of 0.005 at the first analysis, and 0.01 at the second.A specific stopping rule is settled for operative mortality (30 days) at 0.01 at the first interim analysis and 0.05 at the second interim analysis. Given the invasive nature and the costs of the intervention, a stopping rule for futility was settled in case of a lack of difference for the primary outcome. This was settled at a relative risk for the primary outcome not including the hypothesized value of 0.5 within 99% CI at the first interim analysis and 95% CI at the second.

ELIGIBILITY:
Inclusion Criteria:

* Elective CABG operation
* Age > 18 years
* Ejection fraction < 0.35

Exclusion Criteria:

* No consent
* Emergency operation
* Contra-indication to IABP placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Major morbidity according to STS (30-days mortality, mechanical ventilation > 48 hours, mediastinitis, surgical reexploration, stroke, acute renal failure) | 30 days after operation

SECONDARY OUTCOMES:
Time on mechanical ventilation; ICU and hospital stay | 30 days after the operation
IABP complications (lower limb ischemia, mesenteric ischemia, bleeding) | 30 days after the operation

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Policlinico S.Donato, San Donato Milanese, Milan
  - IRCCS Policlinico San Donato, San Donato Milanese (Milan)

REFERENCES:
- [Background] Dyub AM, Whitlock RP, Abouzahr LL, Cina CS. Preoperative intra-aortic balloon pump in patients undergoing coronary bypass surgery: a systematic review and meta-analysis. J Card Surg. 2008 Jan-Feb;23(1):79-86. doi: 10.1111/j.1540-8191.2007.00499.x. PMID 18290898
- [Background] Christenson JT, Licker M, Kalangos A. The role of intra-aortic counterpulsation in high-risk OPCAB surgery: a prospective randomized study. J Card Surg. 2003 Jul-Aug;18(4):286-94. doi: 10.1046/j.1540-8191.2003.02030.x. PMID 12869172
- [Derived] Ranucci M, Castelvecchio S, Biondi A, de Vincentiis C, Ballotta A, Varrica A, Frigiola A, Menicanti L; Surgical and Clinical Outcome Research (SCORE) Group. A randomized controlled trial of preoperative intra-aortic balloon pump in coronary patients with poor left ventricular function undergoing coronary artery bypass surgery*. Crit Care Med. 2013 Nov;41(11):2476-83. doi: 10.1097/CCM.0b013e3182978dfc. PMID 23921278